CLINICAL TRIAL: NCT04345692
Title: A Randomized, Controlled Clinical Trial of the Safety and Efficacy of Hydroxychloroquine for the Treatment of COVID-19 in Hospitalized Patients
Brief Title: A Randomized Controlled Clinical Trial: Hydroxychloroquine for the Treatment of COVID-19 in Hospitalized Patients
Acronym: OAHU-COVID19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: RECOVERY Trial results - no efficacy
Sponsor: Queen's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RA-2020-018
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Randomized, 2 arm, open label hydroxychloroquine plus usual care compared to usual care in hospitalized patients
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydroxychloroquine (Experimental): Hydroxychloroquine 400 mg 2x day by mouth on day 1, followed by 200 mg 2x day by mouth days 2-5
  Interventions: Drug: Hydroxychloroquine
- Usual Care (No Intervention): usual care for hospitalized patients diagnosed with COVID-19

INTERVENTIONS:
Drug: Hydroxychloroquine — oral tablet administered by hospital staff or if discharged before day 5 - self administered oral tablet
  Other Names: Plaquenil
  Arms: Hydroxychloroquine

SUMMARY:
This study is a randomized, open label clinical trial to evaluate the safety and efficacy of hydroxychloroquine (HCQ) plus usual care compared to usual care in approximately 350 hospitalized patients diagnosed with COVID-19. The study will be a 2-arm, non-blinded comparison between open label hydroxychloroquine and usual care. The course of treatment (HCQ) is five days. Participants will be followed to study day 28.

DETAILED DESCRIPTION:
The overall objective is to evaluate the clinical efficacy and safety of hydroxychloroquine (HCQ) relative to standard of care among 350 hospitalized adult patients who have COVID-19.

Primary Aim i. Clinical status (on a 7-point ordinal scale) at day 15

Clinical Status 7-point ordinal scale:

1. Not hospitalized, no limitations on activities
2. Not hospitalized, limitation on activities
3. Hospitalized, not requiring supplemental oxygen
4. Hospitalized, requiring supplemental oxygen
5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
6. Hospitalized, on invasive mechanical ventilation or ECMO
7. Death

After enrollment and randomization there will be baseline and then daily assessments of clinical status and test results and procedures during hospitalization. Course of HCQ treatment is 5 days. Participants are followed daily during hospitalization. All procedures, evaluations and treatment, including the hydroxychloroquine laboratory tests, and radiology tests are part of the usual clinical care for COVID-19 patients. This study will only collect the information obtained as part of hospital standard of care. If the information is not available, it will not be obtained by any other mechanism. After discharge there is a follow up telephone call at day 15 and day 28. Follow-up assessment includes any clinical events, adverse events, and clinic or emergency visits or hospitalizations. Participants in the HCQ arm have safety labs: CBC and Comprehensive Metabolic profile scheduled on day 7 and 14.

ELIGIBILITY:
Inclusion Criteria:

i. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.

ii. Understands and agrees to comply with planned study procedures. iii. Male or female adult ≥18 - 95 years of age at time of enrolment. iv. Laboratory-confirmed SARS-CoV-2 infection in any specimen < 5 days prior to randomization.

v. At least one of the following:

1. Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.) or
2. Clinical assessment (evidence of rales/crackles on exam) AND SpO2 ≤94% on room air vi. Women of childbearing potential must agree to use at least one primary form of contraception for the duration of the study.

Exclusion Criteria:

i. History of liver failure ii. History of stage 4 severe chronic kidney disease or requiring dialysis iii. Self-reported pregnant or breast feeding. iv. Allergy to hydroxychloroquine or choloroquine v. Known contraindication to hydroxychloroquine, including retinopathy, G6PD deficiency, QT prolongation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
i. Clinical status | Clinical Status (on a 7-point ordinal scale) at day 15
  Clinical Status (on a 7-point ordinal scale) at day 15
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities
  3. Hospitalized, not requiring supplemental oxygen
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, on invasive mechanical ventilation or ECMO
  7. Death

SECONDARY OUTCOMES:
Oxygenation | up to day 28
  Oxygenation free days in the first 28 days Incidence and duration of new oxygen use during the study
Mechanical Ventilation | up to day 28
  Ventilator free days in the first 28 days Incidence and duration of new mechanical ventilation use during hospitalization
Hospitalization | up to day 28
  Duration of hospitalization (days)
Mortality | up to day 28
  28-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Todd Seto, MD, Principal Investigator — Queen's Medical Center
Locations (1):
- Queen's Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No